CLINICAL TRIAL: NCT02794571
Title: A Phase Ia/Ib Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of Tiragolumab as a Single Agent and in Combination With Atezolizumab and/or Other Anti-Cancer Therapies in Patients With Locally Advanced or Metastatic Tumors
Brief Title: Safety and Pharmacokinetics (PK) of Escalating Doses of Tiragolumab as a Single Agent and in Combination With Atezolizumab and/or Other Anti-Cancer Therapies in Locally Advanced or Metastatic Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO30103; 2016-000944-33 (EudraCT Number)
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Advanced/Metastatic Tumors
MeSH Terms: conditions — Neoplasm Metastasis | interventions — atezolizumab; Tiragolumab; Carboplatin; Cisplatin; Pemetrexed; Paclitaxel; Etoposide; Capecitabine; Bevacizumab; pembrolizumab

ARMS (12):
- Phase Ia Dose-Escalation Stage: Tiragolumab (Experimental): Cohorts of at least 3 participants each will be treated with escalating doses of tiragolumab.
  Interventions: Drug: Tiragolumab
- Phase Ia Dose-Expansion Stage: Tiragolumab (Experimental): Participants will be treated with tiragolumab at or below the maximum tolerated dose (MTD) or maximum administered dose (MAD) in the study.
  Interventions: Drug: Tiragolumab
- Phase Ib Q3W Dose-Escalation Stage: Tiragolumab+Atezolizumab (Experimental): A minimum of 3 participants will be treated for each dose level of tiragolumab in combination with a fixed dose of atezolizumab with tiragolumab being administered prior to atezolizumab.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Phase Ib Q3W Dose-Expansion Stage: Tiragolumab+Atezolizumab (Experimental): Participants will be treated every 3 weeks (Q3W) with tiragolumab at or below the MTD or MAD in combination with a fixed dose of atezolizumab with tiragolumab being administered prior to atezolizumab.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Phase Ib Chemotherapy Dose-Expansion Stage: Cohort A (Experimental): In Cohort A, carboplatin or cisplatin and pemetrexed chemotherapy will be administered after atezolizumab and tiragolumab intravenous (IV) infusion. During induction phase, participants will receive atezolizumab and tiragolumab in combination with carboplatin or cisplatin and pemetrexed on Day 1 of each 21-day cycle for 4 to 6 cycles. During maintenance phase, participants will receive atezolizumab and tiragolumab in combination with pemetrexed on Day 1 of each 21-day cycle.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed
- Phase Ib Chemotherapy Dose-Expansion Stage: Cohort B (Experimental): In Cohort B, carboplatin and paclitaxel chemotherapy will be administered after atezolizumab and tiragolumab IV infusion. During induction phase, participants will receive atezolizumab and tiragolumab in combination with carboplatin and paclitaxel on Day 1 of each 21-day cycle for 4 to 6 cycles. During maintenance phase, participants will receive atezolizumab and tiragolumab on Day 1 of each 21-day cycle (participants enrolled under protocol version 4) or Day 1 of each 28-day cycle (participants enrolled under protocol version 5).
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Drug: Carboplatin; Drug: Paclitaxel
- Phase Ib Chemotherapy Dose-Expansion Stage: Cohort C (Experimental): In Cohort C, carboplatin or cisplatin and etoposide chemotherapy will be administered after atezolizumab and tiragolumab IV infusion. During induction phase, participants will receive atezolizumab and tiragolumab in combination with carboplatin or cisplatin on Day 1 of each 21-day cycle and etoposide on Day 1 to 3 of each 21-day cycle for 4 cycles. During maintenance phase, participants will receive atezolizumab and tiragolumab on Day 1 of each 28-day cycle.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide
- Phase Ib Chemotherapy Dose-Expansion Stage: Cohort D (Experimental): In Cohort D, participants will receive atezolizumab and tiragolumab on Day 1 and capecitabine on Day 1-14 of each 21-day cycle.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Drug: Capecitabine
- Phase Ib Q4W Sequential Dose-Expansion Stage: Tiragolumab+Atezolizumab (Experimental): Participants will be treated every 4 weeks (Q4W) with fixed doses of tiragolumab and atezolizumab with tiragolumab being administered prior to atezolizumab.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Phase Ib Q4W Coinfusion Expansion Cohort Tiragolumab+Atezolizumab (Experimental): Participants will be treated Q4W with fixed doses of tiragolumab and atezolizumab mixed and administered in one IV bag.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Phase Ib Non-Chemotherapy Dose-Expansion Stage: Cohort NC1 (Experimental): In Cohort NC1, participants will receive atezolizumab and tiragolumab in combination with bevacizumab on Day 1 of each 21-day cycle.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Drug: Bevacizumab
- Phase Ib Non-Chemotherapy Dose-Expansion Stage: Cohort NC2 (Experimental): In Cohort NC2, participants will receive tiragolumab in combination with pembrolizumab on Day 1 of each 21-day cycle.
  Interventions: Drug: Tiragolumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be given as 1200 mg via IV infusion on Day 1 of each 21-day cycle or as 1680 mg via IV infusion on Day 1 of each 28-day cycle.
  Other Names: MPDL3280A; RO5541267; Tecentriq
  Arms: Phase Ib Chemotherapy Dose-Expansion Stage: Cohort A; Phase Ib Chemotherapy Dose-Expansion Stage: Cohort B; Phase Ib Chemotherapy Dose-Expansion Stage: Cohort C; Phase Ib Chemotherapy Dose-Expansion Stage: Cohort D; Phase Ib Non-Chemotherapy Dose-Expansion Stage: Cohort NC1; Phase Ib Q3W Dose-Escalation Stage: Tiragolumab+Atezolizumab; Phase Ib Q3W Dose-Expansion Stage: Tiragolumab+Atezolizumab; Phase Ib Q4W Coinfusion Expansion Cohort Tiragolumab+Atezolizumab; Phase Ib Q4W Sequential Dose-Expansion Stage: Tiragolumab+Atezolizumab
Drug: Tiragolumab — Several dose levels will be evaluated for tiragolumab administered as a single agent and in combination with atezolizumab and/or other anti-cancer therapies. Tiragolumab will be given via IV infusion on Day 1 of each cycle (21-day or 28-day depending on study cohort and phase) until disease progression or loss of clinical benefit. Those who discontinue treatment with single-agent tiragolumab may receive combination treatment with tiragolumab and atezolizumab and/or other anti-cancer therapies. Combination treatment may continue until disease progression or loss of clinical benefit.
  Other Names: MTIG7192A; RO7092284
Drug: Carboplatin — Carboplatin, AUC of 6 milligram per milliliter per minute (mg/ml/min) for Cohorts A and B and AUC of 5 mg/ml/min for Cohort C, IV infusion will be administered on Day 1 of each 21-day cycle after combination treatment of atezolizumab and tiragolumab IV infusion.
  Arms: Phase Ib Chemotherapy Dose-Expansion Stage: Cohort A; Phase Ib Chemotherapy Dose-Expansion Stage: Cohort B; Phase Ib Chemotherapy Dose-Expansion Stage: Cohort C
Drug: Cisplatin — Cisplatin 75 milligram per square meter (mg/m^2) IV infusion will be administered on day 1 of each 21-day cycle after combination treatment of atezolizumab and tiragolumab.
  Arms: Phase Ib Chemotherapy Dose-Expansion Stage: Cohort A; Phase Ib Chemotherapy Dose-Expansion Stage: Cohort C
Drug: Pemetrexed — Pemetrexed 500 mg/m^2 IV infusion will be administered on Day 1 of each 21-day cycle after carboplatin or cisplatin IV infusion with combination treatment of atezolizumab and tiragolumab.
  Arms: Phase Ib Chemotherapy Dose-Expansion Stage: Cohort A
Drug: Paclitaxel — Paclitaxel 200 mg/m^2 IV infusion will be administered on Day 1 of each 21-day cycle after combination treatment with atezolizumab and tiragolumab.
  Arms: Phase Ib Chemotherapy Dose-Expansion Stage: Cohort B
Drug: Etoposide — Etoposide 100 mg/m^2 IV infusion will be administered on Days 1, 2, and 3 of each 21-day cycle with combination treatment of atezolizumab and tiragolumab.
  Arms: Phase Ib Chemotherapy Dose-Expansion Stage: Cohort C
Drug: Capecitabine — Capecitabine 1250 mg/m^2 oral dose will be administered twice daily (BID) on Days 1 through 14 of each 21-day cycle. On Day 1 of Cycle 1, the first dose of capecitabine will be administered prior to the atezolizumab and tiragolumab infusion.
  Arms: Phase Ib Chemotherapy Dose-Expansion Stage: Cohort D
Drug: Bevacizumab — Bevacizumab 15 mg/kg IV infusion will be administered on Day 1 of each 21-day cycle after combination treatment of atezolizumab and tiragolumab.
  Arms: Phase Ib Non-Chemotherapy Dose-Expansion Stage: Cohort NC1
Drug: Pembrolizumab — Pembrolizumab 200 mg IV infusion will be administered on Day 1 of each 21-day cycle after treatment with tiragolumab.
  Arms: Phase Ib Non-Chemotherapy Dose-Expansion Stage: Cohort NC2

SUMMARY:
This first-in-human open-label, multicenter, dose-escalation and expansion study is designed to evaluate the safety, tolerability, and PK of tiragolumab alone or in combination with atezolizumab and/or other anti-cancer therapies in participants with locally advanced, recurrent, or metastatic incurable tumors for whom standard therapy does not exist, has proven to be ineffective or intolerable, or is considered inappropriate, or for whom a clinical trial of an investigational agent is a recognized standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy at least 12 weeks
* Adequate hematologic and end organ function
* Histologic documentation of locally advanced, recurrent, or metastatic incurable malignancy that has progressed after at least one available standard therapy; or for which standard therapy has proven ineffective, intolerable, or considered inappropriate; or for which a clinical trial of an investigational agent is a recognized standard of care
* Confirmed availability of representative tumor specimens
* Measurable disease according to RECIST Version 1.1

Exclusion Criteria:

* Any anti-cancer therapy, whether investigational or approved, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks prior to initiation of study treatment
* Malignancies other than disease under study within 5 years prior to Day 1 of Cycle 1
* Primary central nervous system (CNS) malignancy, or untreated/active CNS metastases
* Leptomeningeal disease
* History of idiopathic pulmonary fibrosis, pneumonitis, organizing pneumonia, or evidence of active pneumonitis on Screening chest computed tomograph (CT) scan
* History of autoimmune disease
* Positive human immunodeficiency virus (HIV) test
* Active hepatitis B or C, or tuberculosis
* Severe infection within 4 weeks prior to randomization
* Prior allogeneic bone marrow or solid organ transplant
* Significant cardiovascular disease
* Known clinically significant liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | From Baseline to the end of Cycle 1 (up to 21 days)
Percentage of Participants with Adverse Events (AEs) Graded per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0 | From Baseline up to 90 days after last dose of study treatment or until initiation of another systemic anti-cancer therapy (up to approximately 8 years)
Number of Cycles with Tiragolumab | From Baseline to last dose (up to approximately 8 years)
Phase Ia and Ib: Percentage of Participants with Anti-Drug Antibodies (ADAs) to Tiragolumab | Day 1 up to 8 years
  Phase (Ph) 1a: Pre-dose on Day 1, Cycles 1-4, 8, 16, every eight cycles (Q8C), at discontinuation (DC), every 30 days up to 120 days (cycle length 21 days); Phase 1b without Chemotherapy: Pre-dose on Day 1, Cycles 1-4, 8, then Q8C, DC (cycle length 21 days); Phase 1b (Chemotherapy Cohorts and Q4W): Pre-dose on Day 1, Cycles 1-4, 8, 12 and 16, then DC (cycle length 21/28 days).
Phase Ib: Percentage of Participants with ADAs to Atezolizumab | Day 1 up to 8 years
  Phase 1b (without Chemotherapy): Pre-dose on Day 1, Cycles 1-4, 8, then Q8C, at DC, every 30 days up to 120 days (cycle length 21 days); Phase 1b (Chemotherapy Cohorts and Q4W): Pre-dose on Day 1, Cycles 1-4, 8, 12 and 16, then DC (cycle length 21/28 days).

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) of Tiragolumab | Day 1 up to 8 years
  During Phase Ia and Phase Ib dose-escalation stages time frame is as follows: Pre-dose Day 1, Cycles 1-4, 8 (cycle length 21 days); Cycle 1: Post-dose-0.5 hour, 24 hours, Days 8 and 15; Day 1, Cycles 2-7 (Ph 1a), Cycles 2, 3, 4 ,8, 16 -0.5 hour post-dose; Ph1a and 1b - Q8C, DC; every 30 days up to 120 days.
  During Phase Ia dose-expansion stage and Phase Ib dose-expansion stages with and without chemotherapy time frame is as follows: Pre-dose Day 1,Cycles 1-4, 8 (cycle length 21/28 days); Cycle 1: Post-dose-0.5 hour, Days 2, 8 and 15 (D2, D8 and D15 only applicable to Q4W co-infusion cohort); Day 1, Cycles 2, 3, 4, 8, 12* 16 (C12* only applicable to Q4W and Chemotherapy cohorts): 0.5 hour post-dose; ph1a and 1b (Q3W)- Q8C, DC; every 30 days up to 120 days.
Maximum Serum Concentration (Cmax) of Tiragolumab | Day 1 up to 8 years
  During Phase Ia and Phase Ib dose-escalation stages time frame is as follows: Pre-dose Day 1,Cycles 1-4, 8 (cycle length 21 days); Cycle 1: Post-dose-0.5 hour, 24 hours, Days 8 and 15; Day 1, Cycles 2-7 (Ph 1a), Cycles 2, 3, 4 ,8, 16 -0.5 h post-dose; ph1a and 1b - Q8C, DC; every 30 days up to 120 days.
  During Phase Ia dose-expansion stage and Phase Ib dose-expansion stages with and without chemotherapy time frame is as follows: Pre-dose Day 1,Cycles 1-4, 8 (cycle length 21/28 days); Cycle 1: Post-dose-0.5 hour, Days 2, 8 and 15 (D2, D8 and D15 only applicable to Q4W co-infusion cohort); Day 1, Cycles 2, 3, 4, 8, 12* 16 (C12* only applicable to Q4W and Chemotherapy cohorts): 0.5 hour post-dose; ph1a and 1b (Q3W)- Q8C, DC; every 30 days up to 120 days.
Minimum Serum Concentration (Cmin) of Tiragolumab | Day 1 up to 8 years
  During Phase Ia and Phase Ib dose-escalation stages time frame is as follows: Pre-dose Day 1,Cycles 1-4, 8 (cycle length 21 days); Cycle 1: Post-dose-0.5 hour, 24 hours, Days 8 and 15; Day 1, Cycles 2-7 (Ph 1a), Cycles 2, 3, 4 ,8, 16 -0.5 hour post-dose; ph1a and 1b - Q8C, DC; every 30 days up to 120 days.
  During Phase Ia dose-expansion stage and Phase Ib dose-expansion stages with and without chemotherapy time frame is as follows: Pre-dose Day 1,Cycles 1-4, 8 (cycle length 21/28 days); Cycle 1: Post-dose-0.5 hour, Days 2, 8 and 15 (D2, D8 and D15 only applicable to Q4W co-infusion cohort); Day 1, Cycles 2, 3, 4, 8, 12* 16 (C12* only applicable to Q4W and Chemotherapy cohorts): 0.5 h post-dose; ph1a and 1b (Q3W)- Q8C, DC; every 30 days up to 120 days.
Clearance (CL) of Tiragolumab | Day 1 up to 8 years
  During Phase Ia and Phase Ib dose-escalation stages time frame is as follows: Pre-dose Day 1,Cycles 1-4, 8 (cycle length 21 days); Cycle 1: Post-dose-0.5 hour, 24 hours, Days 8 and 15; Day 1, Cycles 2-7 (Ph 1a), Cycles 2, 3, 4 ,8, 16 -0.5 hour post-dose; ph1a and 1b - Q8C, DC; every 30 days up to 120 days.
  During Phase Ia dose-expansion stage and Phase Ib dose-expansion stages with and without chemotherapy time frame is as follows: Pre-dose Day 1,Cycles 1-4, 8 (cycle length 21/28 days); Cycle 1: Post-dose-0.5 hour, Days 2, 8 and 15 (D2, D8 and D15 only applicable to Q4W co-infusion cohort); Day 1, Cycles 2, 3, 4, 8, 12* 16 (C12* only applicable to Q4W and Chemotherapy cohorts): 0.5 hour post-dose; ph1a and 1b (Q3W)- Q8C, DC; every 30 days up to 120 days.
Volume of Distribution at Steady State (Vss) of Tiragolumab | Day 1 up to 8 years
  During Phase Ia and Phase Ib dose-escalation stages time frame is as follows: Pre-dose Day 1,Cycles 1-4, 8 (cycle length 21 days); Cycle 1: Post-dose-0.5 hour, 24 hours, Days 8 and 15; Day 1, Cycles 2-7 (Ph 1a), Cycles 2, 3, 4 ,8, 16 -0.5 hour post-dose; ph1a and 1b - Q8C, DC; every 30 days up to 120 days.
  During Phase Ia dose-expansion stage and Phase Ib dose-expansion stages with and without chemotherapy time frame is as follows: Pre-dose Day 1, Cycles 1-4, 8 (cycle length 21/28 days); Cycle 1: Post-dose-0.5 hour, Days 2, 8 and 15 (D2, D8 and D15 only applicable to Q4W co-infusion cohort); Day 1, Cycles 2, 3, 4, 8, 12* 16 (C12* only applicable to Q4W and Chemotherapy cohorts): 0.5 hour post-dose; ph1a and 1b (Q3W)- Q8C, DC; every 30 days up to 120 days.
Cmax of Atezolizumab | Day 1 up to 8 years
  During Phase Ib dose-escalation stage time frame will be as follows: Pre-dose Day 1,Cycles 1-4, 8 (cycle length 21 days); Cycle 1: Post-dose-0.5 hour, 24 hours, Days 8 and 15; Day 1, Cycles 2 ,3, 4, 8, 16: 0.5 hour post-dose; Q8C, DC; every 30 days up to 120 days.
  During Phase Ib dose-expansion stages time frame will be as follows: Pre-dose on Day 1 of Cycles (cycle length 21/28 days) 1-4, 8, 12*, 16 (C12* only applicable to Q4W and Chemotherapy cohorts); Post-dose 0.5 hour on Day 1 of Cycles 1-4, 8, 12, 16; then Q8C until/at DC, every 30 days up to 120 days. For Q4W co-infusion cohort only: post-dose Days 2, 8 and 15 of Cycle 1.
Cmin of Atezolizumab | Day 1 up to 8 years
  During Phase Ib dose-escalation stage time frame will be as follows: Pre-dose Day 1, Cycles 1-4, 8 (cycle length 21 days); Cycle 1: Post-dose-0.5 hour, 24 hours, Days 8 and 15; Day 1, Cycles 2 ,3, 4, 8, 16: 0.5 hour post-dose; Q8C, DC; every 30 days up to 120 days.
  During Phase Ib dose-expansion stages time frame will be as follows: Pre-dose on Day 1 of Cycles (cycle length 21/28 days) 1-4,8, 12*, 16 (C12* only applicable to Q4W and Chemotherapy cohorts); Post-dose 0.5 hour on Day 1 of Cycles 1-4, 8, 12, 16; then Q8C until/at DC, every 30 days up to 120 days. For Q4W co-infusion cohort only: post-dose Days 2, 8 and 15 of Cycle 1.
Plasma Concentration of Cisplatin | Pre-dose (5 min) and post-dose (1 hour) on Day 1 of Cycles 1 and 3 (cycle length 21 days)
Plasma Concentration of Carboplatin | Pre-dose (5 min) and post-dose (1 hour) on Day 1 of Cycles 1 and 3 (cycle length 21 days)
Plasma Concentration of Pemetrexed | Pre-dose (5 min) and post-dose (1 hour) on Day 1 of Cycles 1 and 3 (cycle length 21 days)
Plasma Concentration of Paclitaxel | Pre-dose (5 min) and post-dose (1 hour) on Day 1 of Cycles 1 and 3 (cycle length 21 days)
Plasma Concentration of Etoposide | Pre-dose (5 min) and post-dose (1 hour) on Day 1 of Cycles 1 and 3 (cycle length 21 days)
Plasma Concentration of Capecitabine | Pre-dose (5 min) on Day 1 of Cycle 1 and post-dose (2 hours) on Day 1 of Cycle 3 (cycle length 21 days)
Objective Response According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | From Baseline until disease progression (up to 8 years)
Duration of Objective Response (DOR) According to RECIST Version 1.1 | From Baseline until disease progression (up to 8 years)
Progression-Free Survival (PFS) According to RECIST Version 1.1 | From Baseline until disease progression (up to 8 years)
Overall survival (OS) According to RECIST Version 1.1 | Baseline until death from any cause (up to approximately 8 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (28):
- United States (8):
  - Honor Health Research Institute, Scottsdale, Arizona
  - University of California Los Angeles, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Tennessee Oncology - Nashville, Nashville, Tennessee
- Australia (2):
  - Kinghorn Cancer Centre; St Vincents Hospital, Darlinghurst, New South Wales
  - Peter MacCallum Cancer Center, North Melbourne, Victoria
- Princess Margaret Hospital, Toronto, Ontario, Canada
- France (5):
  - Institut Bergonie CLCC Bordeaux, Bordeaux
  - Centre Léon Bérard Centre Régional de Lutte Contre Le Cancer Rhône Alpes, Lyon
  - Institut Curie, Paris
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Institut Gustave Roussy, Villejuif
- Japan (2):
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Tokyo
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - ICO L'Hospitalet; Servicio de oncologia medica, L'Hospitalet de Llobregat, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Sant Andreu de la Barca, Barcelona
  - Clinica Universitaria de Navarra; Servicio de oncología, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Hospital Universitario HM Sanchinarro-CIOCC; Oncología Médica, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Shemesh CS, Wang Y, An A, Ding H, Chan P, Liu Q, Chen YW, Wu B, Wu Q, Wang X. Phase I pharmacokinetic, safety, and preliminary efficacy study of tiragolumab in combination with atezolizumab in Chinese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2024 Jul;94(1):45-55. doi: 10.1007/s00280-024-04650-y. Epub 2024 Mar 7. PMID 38451273
- [Derived] Garralda E, Oh DY, Italiano A, Bedard PL, Delord JP, Calvo E, LoRusso P, Wainberg Z, Cervantes A, Rodriguez-Vida A, Shemesh CS, Sane R, Mendus D, Ding H, Hendricks R, Meng R, Cho BC, Kim TW, Wu B. Pharmacokinetics (PK) of Tiragolumab in First-in-Human Study in Patients with Mixed Solid Tumors (GO30103). J Clin Pharmacol. 2024 May;64(5):544-554. doi: 10.1002/jcph.2397. Epub 2024 Jan 17. PMID 38105505
- [Derived] Kim TW, Bedard PL, LoRusso P, Gordon MS, Bendell J, Oh DY, Ahn MJ, Garralda E, D'Angelo SP, Desai J, Hodi FS, Wainberg Z, Delord JP, Cassier PA, Cervantes A, Gil-Martin M, Wu B, Patil NS, Jin Y, Hoang T, Mendus D, Wen X, Meng R, Cho BC. Anti-TIGIT Antibody Tiragolumab Alone or With Atezolizumab in Patients With Advanced Solid Tumors: A Phase 1a/1b Nonrandomized Controlled Trial. JAMA Oncol. 2023 Nov 1;9(11):1574-1582. doi: 10.1001/jamaoncol.2023.3867. PMID 37768658